CLINICAL TRIAL: NCT02257476
Title: A Phase I Study of Extended Infusion Carfilzomib on a Weekly Schedule in Patients With Advanced Solid Malignancies
Brief Title: Extended Infusion Carfilzomib on a Weekly Schedule in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, Bradley Carthon MD, PhD, Assistant Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00071307; WINSHIP2598-13 (Other: Winship Cancer Institute)
Record Dates: First submitted 2014-09-26; First posted 2014-10-06 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Neoplasms; Malignancies
Keywords: carfilzomib; advanced solid malignancies; advanced solid cancers; prostate; bladder; colon; breast; lung
MeSH Terms: conditions — Neoplasms | interventions — carfilzomib; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Carfilzomib (Experimental): Patients will receive single agent carfilzomib on a weekly dosing schedule (days 1, 8, 15) in a 21 day cycle. The initial dose will be 20 mg/m² for cycle 1, day 1. Dose escalation will proceed in a standard 3+3 fashion with the requirement that dose escalation to the next level can only proceed if 0 of 3 or ≤ 1 of 6 patients experience a dose limiting toxicity (DLT). Dexamethasone 8 mg PO/IV will be administered prior to all carfilzomib doses.
  Interventions: Drug: Carfilzomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Carfilzomib — Carfilzomib will be given as an IV infusion over 4 hours. Subjects will remain at the clinic under observation for at least 1 hour following each dose of carfilzomib in Cycle 1 and following the dose on Cycle 2 Day 1. During these observation times, post dose IV hydration may be given at physician's discretion.
  Other Names: PR-171; Kyprolis
Drug: Dexamethasone — Dexamethasone 8 mg PO/IV will be administered prior to all carfilzomib doses.
  Other Names: Decadron

SUMMARY:
The purpose of this study is to find the safest dose level of an approved drug, carfilzomib, in solid tumors when given over a different period of time than normally used. The study will also use markers in blood from routine blood draws to help check the levels of the drug. Lastly, the study will check how well this drug works with regards to keeping cancer cells from growing with the new time frame of delivery.

DETAILED DESCRIPTION:
The role of the proteasome in carcinogenesis and cell survival has been well established, and its inhibition associated with an accumulation of pro-apoptotic proteins and cell death. Proteasome inhibitors, such has bortezomib, have been extensively studied and are widely used as effective therapy in the treatment for hematologic malignancies, such as multiple myeloma where circulating proteasome levels have been correlated with survival. Carfilzomib, a novel irreversible proteasome inhibitor which specifically targets the chymotryptic site of the proteasome has shown more potency than bortezomib and may be able to overcome bortezomib resistance. Response rates between 25-54% were seen in patients with previously treated myeloma in the phase 2 setting.

Given the effectiveness of proteasome inhibition in multiple myeloma, the role of proteasome in solid tumors is under active investigation. Previous trials of bortezomib in breast, prostate, lung, and pancreatic cancer have shown little activity of this agent in these diseases. Whether the lack of activity may be mechanistically related (bortezomib inhibits chymotrypsin-like and peptidyl-glutamyl peptide-hydrolyzing (PGPH)-like activities of the proteasome), or a lack of potency in target inhibition, is unknown.

In a phase Ib/II study of 14 patients (phase I) and 51 patients (phase II) with advanced solid tumors, Rosen and colleagues noted single-agent activity with carfilzomib. Carfilzomib was dosed on days 1, 2, 8, 9, 15, and 16 of a 28 day cycle to a maximum of 12 cycles, with 20-36 mg/m² noted as the recommended phase 2 dose based on DLT data. A PR in both renal and small cell lung cancer, and stable disease > 16 weeks in mesothelioma, ovarian, renal, and non-small cell lung cancer was observed. The treatment was tolerable with the most common adverse events (AEs) including fatigue, headache, diarrhea, nausea and constipation.

Given the activity of carfilzomib seen in selected solid tumors, and unpublished data to suggest weekly dosing may result in a similar pharmacokinetic profile including AUC, the investigators propose to study the safety, tolerability, pharmacokinetics, and anti-tumor activity of carfilzomib monotherapy given on a weekly dosing schedule. Weekly dosing has the advantage of patient convenience, and if acceptable toxicity and pharmacokinetics, it allows for easier integration of this schedule into subsequent combination therapy clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years or older at the time of enrollment.
* Advanced/metastatic solid tumor refractory to standard therapy.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 - 2.
* Adequate organ function as assessed by the following:

  * Bone marrow:

    * Hemoglobin greater than or equal to 9.0 g/dL
    * Absolute neutrophil count (ANC) greater than or equal to 1,500/mm³
    * Platelet count greater than or equal to 100,000/mm³
  * Hepatic:

    * Total bilirubin less than or equal to 1.5 x ULN
    * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 3 x ULN
    * Prothrombin time (PT)-international normalized ratio (INR)/partial thromboplastin time (PTT) < 1.5 x ULN except in patients receiving active anticoagulation
  * Renal:

    * Serum creatinine ≤ 1.5 x upper limit of normal or
    * Glomerular filtration rate (GFR) of 50 ml/minute or greater (if elevated serum creatinine level > 1.5 x ULN)
* Willingness to sign informed consent by patient or patient's legal representative.
* Patient with known but adequately treated brain metastases and without central nervous system (CNS) disease progression as determined by CT or MRI imaging within 4 weeks of the first dose of study drug.

Exclusion Criteria:

* Treatment related residual toxicity > grade 1.
* Prior treatment with a proteasome inhibitor.
* Uncontrolled systemic disease or intercurrent illness.
* Recent history of myocardial infarction (MI) or symptomatic coronary artery disease within the preceding 6 months.
* History of uncontrolled hypertension (systolic > 150 mmHg or diastolic pressure > 90 mmHG despite optimal medical management).
* Ejection fraction < 50%.
* Known and actively treated infection with human immunodeficiency virus (HIV), hepatitis B or C.
* Major surgery or significant traumatic injury within 4 weeks of first study treatment from which the subject has not fully recovered.
* Pregnant or breast feeding women.
* Female patient of child-bearing potential or male patient with partner of child-bearing potential but unable or unwilling to use effective contraception (double barrier such as condoms, contraceptive sponge, diaphragm or vaginal ring with spermicidal jellies or cream; or hormonal method such as oral, parenteral or transdermal hormonal agents for at least three months prior to study drug administration).
* Corticosteroid doses greater than equivalent of prednisone 7.5 mg PO daily.
* Recent therapy with any active anticancer agent within 4 weeks of the 1st dose of the study drugs.
* Any other current malignancy or previous malignancies within 3 years of enrollment except: curatively treated in situ carcinoma of the cervix uteri; localized basal or squamous cell carcinoma of the skin, curatively treated in situ breast carcinoma, and early stage prostate cancer.
* Known history of allergy to Captisol® (a cyclodextrin derivative used to solubilize carfilzomib).
* Contraindication to any of the required concomitant drugs or supportive treatments, including hypersensitivity to all anticoagulation and antiplatelet options, antiviral drugs, or intolerance to hydration due to preexisting pulmonary or cardiac impairment.
* Subjects with pleural effusions requiring thoracentesis or ascites requiring paracentesis within 14 days prior to randomization.
* Any other clinically significant medical disease or condition that, in the Investigator's opinion, may interfere with protocol adherence or a subject's ability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) of a weekly 4-hour carfilzomib infusion in patients with advanced solid malignancies | Up to 18 months
  Evaluate safety and tolerability of weekly dosed carfilzomib as assessed by using NCI Common Toxicity Criteria for Adverse Effects (CTCAE) v.4 criteria to determine DLTs, the MTD, and RP2D

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of escalating doses of weekly intravenous carfilzomib | 1, 2, 4, 6, 8, 28 hours post-dose
  Pharmacokinetic analysis (Tmax, Cmax, t1/2, AUC)
Changes in pharmacodynamic (PD) biomarkers before and during treatment with carfilzomib using peripheral blood mononuclear cells (PBMC) and paired tumor biopsies | Days 1, 2, 3, 8, 15, 21
  Pharmacodynamic (PD) evaluation of degree of 20S proteasomal inhibition in PBMC assays conducted at Emory University before treatment and at time of first restaging scan
Preliminary anti-tumor efficacy (objective response rate) | Up to 18 months
  Objective Response Rate (CR + PR) by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria in patients who completed at least 2 cycles of protocol therapy
Preliminary anti-tumor efficacy (clinical benefit rate) | Up to 18 months
  Clinical Benefit Rate (CR + PR + SD) by RECIST 1.1 criteria in patients who completed at least 2 cycles of protocol therapy
Preliminary anti-tumor efficacy (progression free survival) | Up to 18 months
Preliminary anti-tumor efficacy (overall survival) | Up to 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Bradley C. Carthon, MD, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University Winship Cancer Institute, Atlanta, Georgia, United States